CLINICAL TRIAL: NCT01125007
Title: Biofilm Capacity Removal and Gingival Abrasion After Utilization Medium and Soft Toothbrushes
Brief Title: Capacity of Biofilm Removal and Gingival Abrasion After Utilization Medium and Soft Toothbrushes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Franciscan University Center (Other)
Responsible Party: Ana Maria Chagas, coordinator
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: FranciscanUC
Record Dates: First submitted 2010-05-14; First posted 2010-05-18 (Estimated); Last update posted 2010-05-18 (Estimated); Status verified 2009-01

CONDITIONS: Biofilm Removal; Gingival Abrasion
Keywords: Dental plaque; Gingival abrasion; toothbrushing
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- toothbrush (Active Comparator): a randomization was performed in which the participants were allocated to the following experimental procedures: Two quadrants (1 and 3 or 2 and 4) with medium toothbrush Two quadrants with soft toothbrush. All procedures were performed using the same dentifrice. Each quadrant was brushed for 30 seconds by the participant without specific instructions on the technique, under supervision of the person in charge of the randomization.
  Interventions: Device: Two kind toothbrushes
- medium toothbrush (Experimental): a randomization was performed in which the participants were allocated to the following experimental procedures: Two quadrants (1 and 3 or 2 and 4) with medium toothbrush Two quadrants with soft toothbrush. All procedures were performed using the same dentifrice. Each quadrant was brushed for 30 seconds by the participant without specific instructions on the technique, under supervision of the person in charge of the randomization.
  Interventions: Device: Two kind toothbrushes

INTERVENTIONS:
Device: Two kind toothbrushes — a randomization was performed in which the participants were allocated to the following experimental procedures: Two quadrants (1 and 3 or 2 and 4) with medium toothbrush Two quadrants with soft toothbrush. All procedures were performed using the same dentifrice. Each quadrant was brushed for 30 seconds by the participant without specific instructions on the technique, under supervision of the person in charge of the randomization.

SUMMARY:
This study compared the removal of dental biofilm between soft and medium toothbrushes. The patients refrained from performing mechanical or chemical plaque control for 96 hours to allow dental biofilm accumulation on the tooth surfaces. After the period of dental biofilm formation, the quadrants were randomized and the participants brushed different quadrants with soft and medium toothbrushes, with or without dentifrice. The plaque indices were analyzed by a blinded examiner before and after toothbrushing. The 2Tone was used for plaque disclosure and analysis was performed by the Quigley-Hein index modified by Turesky et al. (1970).

ELIGIBILITY:
Inclusion Criteria:

* The study was conducted on 25 participants selected among undergraduate dental students of UNIFRA (Santa Maria, Rio Grande do Sul, Brazil)
* Males and Females
* All systemically healthy
* Aged 18 to 30 years (mean age 21.4 ± 3.9 years) with at least 20 present teeth

Exclusion Criteria:

* The exclusion criteria comprised presence of sites with attachment loss ≥ 2mm
* Orthodontic appliances
* Prostheses
* Dental implants
* Aabrasions, restorations and/or carious lesions on the cervical region

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2009-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Gingival abrasion | Presence of gingival abrasion
  All gingival quadrants were analised by photographs made in different experimental times. After that, all photographs were evaluated in a blinded manner, according to the methodology suggested by Danser, et al. (1998), dividing the region to be analyzed in three areas: cervical, interdental and mid-gingival. In each area, the presence of gingival abrasion was assessed dichotomically.

CONTACTS AND LOCATIONS:
Locations (1):
- Franciscan Universtity center, Santa Maria, Rio Grande do Sul, Brazil